CLINICAL TRIAL: NCT01285999
Title: PLATINUM China: A Prospective, Randomized, Multicenter Trial to Assess an Everolimus-Eluting Coronary Stent System (PROMUS™ Element™) for the Treatment of a Single De Novo Coronary Artery Lesion
Brief Title: Prospective, Randomized, Multicenter Trial to Assess PROMUS™ Element™ Stent
Acronym: PTChina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2227
Record Dates: First submitted 2011-01-25; First posted 2011-01-31 (Estimated); Results first posted 2024-11-20 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Atherosclerosis; Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROMUS Element (Experimental): PROMUS Element Everolimus-Eluting Coronary Stent System (PROMUS Element)
  Interventions: Device: PROMUS Element Coronary Stent System
- TAXUS Liberté DES (Active Comparator): TAXUS Liberté Paclitaxel-Eluting Coronary Stent System (TAXUS Liberté)
  Interventions: Device: TAXUS Liberté Coronary Stent System

INTERVENTIONS:
Device: PROMUS Element Coronary Stent System — Everolimus-eluting Coronary Stent Drug-eluting Stent (DES) implantation
  Arms: PROMUS Element
Device: TAXUS Liberté Coronary Stent System — Paclitaxel-eluting Coronary Stent Drug-eluting Stent (DES) implantation
  Arms: TAXUS Liberté DES

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the PROMUS™ Element™ Everolimus-Eluting Coronary Stent System for the treatment of subjects in China with a single de novo atherosclerotic coronary artery lesion.

DETAILED DESCRIPTION:
A prospective, multi-center, randomized-controlled, single-blind, superiority trial at up to 15 sites in China to enroll 500 subjects (3:1 randomization PROMUS Element to TAXUS Liberté) with a single de novo lesion <38mm in length (by visual estimate) in a native coronary artery ≥2.50mm to ≤4.00 mm in diameter (by visual estimate).

ELIGIBILITY:
Clinical Inclusion Criteria:

* Subject must be age 18 - 75 years
* Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial- specific tests or procedures are performed
* Subject is eligible for percutaneous coronary intervention (PCI)
* Subject has symptomatic coronary artery disease or documented silent ischemia
* Subject is an acceptable candidate for coronary artery bypass grafting (CABG)
* Subject has a left ventricular ejection fraction (LVEF) ≥30% as measured within 60 days prior to enrollment
* Subject is willing to comply with all protocol-required follow-up evaluations

Angiographic Inclusion Criteria:

* Target lesion must be a de novo lesion located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥2.50 mm and ≤ 4.00 mm.
* Target lesion length must measure <38 mm (by visual estimate)
* Target lesion must have visually estimated stenosis ≥50% and <100% with Thrombolysis in Myocardial Infarction (TIMI) flow >1.
* Target lesion must be successfully pre-dilated.

Exclusion Criteria:

* Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute MI
* Subject with unstable angina or recent MI (within 1 week) must have creatine kinase (CK)/ creatine kinase-myoglobin band(CK-MB) or troponin documented prior to the procedure and are excluded if any of the following criteria are met at the time of the index procedure:

  * of CK MB >2× upper limit of normal (ULN), the subject is excluded regardless of the CK Total.
  * If CK Total >2× ULN, either CK-MB or troponin must be drawn and the subject is excluded if either CK-MB or troponin is abnormal.
  * If neither CK Total or CK MB is drawn but troponin is, the subject is excluded if troponin >1× ULN and the subject has at least one of the following:

    * Subject has ischemic symptoms and ECG changes indicative of ongoing ischemia (e.g., >1 mm stent thrombosis (ST) segment elevation or depression in consecutive leads or new left bundle branch block (LBBB)
    * Development of pathological Q waves in the ECG or;
    * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality Note: Subjects who do not have recent MI or unstable angina must still have CK/CK-MB or troponin drawn prior to the index procedure. However, the results for these subjects do not need to be available prior to the index procedure and there are no exclusion criteria based on these laboratory studies.
* Subject has received an organ transplant or is on a waiting list for an organ transplant
* Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* Subject is receiving oral or intravenous immunosuppressive therapy (Note: use of inhaled steroids does not exclude subjects) or has known life- limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus; Note: this does not include diabetes mellitus)
* Subject is receiving chronic (≥72 hours) anticoagulation therapy (e.g., heparin, coumadin) for indications other than acute coronary syndrome
* Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Subject has a white blood cell (WBC) count <3,000 cells/mm3
* Subject has documented or suspected liver disease, including laboratory evidence of hepatitis
* Subject is on dialysis or has serum creatinine level >2.0 mg/dL
* Subject has active peptic ulcer disease, an active gastrointestinal (GI) bleed, other bleeding diathesis or coagulopathy or will refuse transfusions
* Subject has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months, or has any permanent neurologic defect that may cause non-compliance with the protocol
* Target vessel (including side branches) has been treated with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) within 12 months prior to the index procedure
* Target vessel has been treated within 10 mm proximal or distal to the target lesion (by visual estimate) with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) at any time prior to the index procedure
* Non-target vessel has been treated with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) within 24 hours prior to the index procedure
* Planned or actual target vessel treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon, or transluminal extraction catheter immediately prior to stent placement
* Planned PCI or CABG after the index procedure
* Subject previously treated at any time with coronary intravascular brachytherapy
* Subject has known allergy to the study stent system or protocol-required concomitant medications (e.g., everolimus, paclitaxel or structurally related compounds; fluoropolymers; thienopyridines or aspirin; contrast; acrylic; stainless steel; platinum; chromium; nickel; iron; tungsten) that cannot be adequately premedicated
* Subject has any other serious medical illness (e.g., cancer, congestive heart failure) that may reduce life expectancy to less than 12 months
* Subject has current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.)
* Subject has a planned procedure that may cause non-compliance with the protocol or confound data interpretation
* Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint or intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
* Subject with known intention to procreate within 12 month after the index procedure (Women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 month after the index procedure.)
* Subject is a woman who is pregnant or nursing (A pregnancy test must be performed within 7 days prior to the index procedure in women of child- bearing potential.)
* Subject has more than 1 lesion that requires treatment during the index procedure

Angiographic Exclusion Criteria:

* Target lesion meets any of the following criteria:

  * Left main location
  * Located within 5 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCX) coronary artery or Right Coronary Artery (RCA) by visual estimate
  * Located within a saphenous vein graft or an arterial graft
  * Will be accessed via a saphenous vein graft or an arterial graft
  * Involves a side branch ≥2.0 mm in diameter by visual estimate
  * Involves a side branch <2.0 mm in diameter by visual estimate which requires treatment
  * TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
  * Excessive tortuosity proximal to or within the lesion
  * Excessive angulation proximal to or within the lesion
  * Target lesion and/or target vessel proximal to the target lesion is moderately to severely calcified by visual estimate
  * Restenotic from previous intervention
  * Thrombus, or possible thrombus, present in the target vessel
  * Target lesion cannot be covered by a single study stent (unplanned bailout stenting is allowed)
* Subject has unprotected left main coronary artery disease (>50% diameter stenosis)
* Subject has protected left main coronary artery disease (>50% diameter stenosis in the left main coronary artery (LMCA) with bypass graft[s] to the left coronary artery) and a target lesion in the LAD or LCX
* Subject has an additional clinically significant lesion(s) for which an intervention within 12 months after the index procedure may be required

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuejin Yang, Principal Investigator — Cardiovascular Institute and Fu Wai Hospital
Locations (15):
- China (15):
  - Cardiovascular Institute and Fu Wai Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - The Chinese People's Liberation Army General Hospital, Beijing
  - Huaxi Hospital of Sichuan University, Chengdu
  - Daqing General Oil Field Hospital, Daqing
  - Guangdong Cardiovascular Institute of Guangdong Provincial Hospital, Guangzhou
  - Guangdong Nanfang Hospital, Guangzhou
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin
  - Nanjing First Hospital, Nanjing
  - Shanghai 6th People's Hospital, Jiaotong University, Shanghai
  - Shanghai Chest Hospital of Jiaotong University, Shanghai
  - General Hospital of SY Military Institute, Shenyang
  - TEDA International Cardiovascular Hospital, Tianjin
  - Xijing Hospital, Fourth Military Medical University, Xi'an

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao R, Han Y, Yang Y, Zhang J, Hou Y, Wang H, Li H, Fang Q, Yu B, Xu B, Allocco DJ, Dawkins KD. PLATINUM China: a prospective, randomized investigation of the platinum chromium everolimus-eluting stent in de novo coronary artery lesions. Catheter Cardiovasc Interv. 2015 Mar;85 Suppl 1:716-23. doi: 10.1002/ccd.25859. Epub 2015 Feb 18. PMID 25631909

RESULTS

PARTICIPANT FLOW:
Groups:
- TAXUS Liberté DES: TAXUS Liberté Paclitaxel-Eluting Coronary Stent System (TAXUS Liberté)
  TAXUS Liberté Coronary Stent System: Paclitaxel-eluting Coronary Stent Drug Eluting Stent (DES) implantation
Period: Overall Study
Arm/Group | PROMUS Element | TAXUS Liberté DES
Started | 373 | 127
Completed | 373 | 127
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PROMUS Element: PROMUS Element Everolimus-Eluting Coronary Stent System (PROMUS Element)
  PROMUS Element Coronary Stent System: Everolimus-eluting Coronary Stent DES implantation
- TAXUS Liberté DES: TAXUS Liberté Paclitaxel-Eluting Coronary Stent System (TAXUS Liberté)
  TAXUS Liberté Coronary Stent System: Paclitaxel-eluting Coronary Stent DES implantation
- Total: Total of all reporting groups
Arm/Group | PROMUS Element | TAXUS Liberté DES | Total
Number analyzed (Participants) | 373 | 127 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.12 (9.90) | 57.55 (9.50) | 57.23 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 39 | 144
  Male | 268 | 88 | 356
Region of Enrollment [Number; unit: participants]
  China | 373 | 127 | 500

OUTCOME MEASURES:

1. Primary Outcome: 9 Month In-stent Late Loss
Description: The primary endpoint is in-stent late loss measured by quantitative coronary angiography (QCA) at 9 months post-index procedure.
Time Frame: 9 Months
Measure: Number; unit: percentage of Intent-to-treat patients
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of Intent-to-treat patients | 0.11 | 0.40
Statistical Analysis 1: Comparison: PROMUS Element vs TAXUS Liberté DES; H0: μt - μc = 0 H1: μt - μc ≠ 0 where μt and μc are the mean 9-month in-stent late loss values for the subjects in the PROMUS Element test and TAXUS Liberté control treatment groups, respectively; Test type: Superiority or Other; p = 0.05, t-test, 2 sided — p-value has not been adjusted; No adjustment; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.37 to -0.21]

2. Secondary Outcome: Target Vessel Failure (TVF) Rate
Time Frame: In hospital and at 2 years
Population: Per Protocol Population
Measure: Number; unit: percentage of participant
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participant | 3.0 | 5.5

3. Secondary Outcome: Target Lesion Revascularization (TLR) Rate
Time Frame: In hospital and at 2 years
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants | 2.4 | 4.7

4. Secondary Outcome: Target Vessel Revascularization (TVR) Rate
Time Frame: In hospital and at 2 years
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants | 3.0 | 5.5

5. Secondary Outcome: Target Lesion Failure (TLF) Rate
Time Frame: In hospital and at 2 years
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants | 2.4 | 4.7

6. Secondary Outcome: Major Adverse Cardiac Event (MACE) Rate
Time Frame: In hospital and at 2 years
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants | 3.0 | 7.1

7. Secondary Outcome: Myocardial Infarction (MI)(Q-wave and Non-Q-wave) Rate
Time Frame: In hospital and at 2 years
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants | 0.3 | 1.6

8. Secondary Outcome: Cardiac Death Rate
Time Frame: In hospital and at 2 years
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants | 0 | 0

9. Secondary Outcome: Non-cardiac Death Rate
Time Frame: In hospital and at 2 years
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants | 0.0 | 1.6

10. Secondary Outcome: All Death Rate
Time Frame: In hospital and at 2 years
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants | 0.0 | 1.6

11. Secondary Outcome: Cardiac Death or MI Rate
Time Frame: In hospital and at 2 years
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants | 0.3 | 3.1

12. Secondary Outcome: Stent Thrombosis Rate (Definite or Probable by Academic Research Consortium [ARC] Definitions)
Time Frame: In hospital and at 2 years
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants | 0.3 | 0.8

13. Secondary Outcome: Angiographic Endpoints: In-stent and In-segment Percent Diameter Stenosis (%DS), In-segment Late Loss , In-stent and In-segment Minimum Lumen Diameter (MLD)
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage
  In-stent percent diameter stenosis | 11.06 (13.86) | 22.20 (16.00)
  in-segment percent diameter stenosis | 21.51 (12.17) | 28.42 (14.92)
  In-segment late loss | 0.06 (0.36) | 0.27 (0.45)
  In-stent minimum lumen diameter | 2.52 (0.53) | 2.24 (0.57)
  in-segment minimum lumen diameter | 2.24 (0.52) | 2.07 (0.56)

14. Secondary Outcome: Periprocedural Endpoints: Technical Success Rate, Clinical Procedural Success Rate
Time Frame: In hospital
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants
  Technical success rate | 99.5 | 99.2
  Clinical procedural success rate | 100.00 | 100.00

15. Secondary Outcome: Angiographic Endpoints: In-stent and In-segment Binary Restenosis Rate, Stent Fracture Rate
Time Frame: 9 month
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
percentage of participants
  In-stent binary restenosis rate | 2.1 | 5.2
  in-segment binary restenosis rate | 3.0 | 7.8
  Stent fracture rate | 0.0 | 0.0

16. Secondary Outcome: Minimal Lumen Diameter (QCA), Acute Gain (QCA)
Time Frame: In hospital
Measure: Number; unit: mm
Arm/Group | PROMUS Element | TAXUS Liberté DES
Number analyzed (Participants) | 373 | 127
mm
  In-Stent MLD | 2.64 | 2.65
  Proximal Edge MLD | 2.84 | 2.94
  Distal Edge MLD | 2.44 | 2.43
  In-Stent Acute gain (QCA) | 1.73 | 1.77
  In Segment Acute gain (QCA) | 1.41 | 1.46

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | PROMUS Element | TAXUS Liberté DES
Serious Adverse Events (participants affected / at risk) | 57/373 | 23/127
Other Adverse Events (participants affected / at risk) | 86/373 | 28/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS Element (N=373) | TAXUS Liberté DES (N=127)
Angina pectoris (Cardiac disorders) | 9 (11) | 5 (7)
Angina unstable (Cardiac disorders) | 10 (10) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 8 (9) | 5 (5)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 8 (8) | 1 (2)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arteriosclerosis obliterans (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS Element (N=373) | TAXUS Liberté DES (N=127)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 4 (5) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 4 (4)
Myocardial infarction (Cardiac disorders) | 20 (20) | 9 (9)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 11 (11) | 3 (3)
Non-cardiac chest pain (General disorders) | 7 (7) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Troponin I increased (Investigations) | 5 (5) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No